CLINICAL TRIAL: NCT04867525
Title: Clinical Research Platform for Molecular Testing, Treatment, Quality of Life and Outcome of Patients With Metastatic Colorectal Cancer Receiving Systemic Therapy (AZURITE)
Brief Title: Registry Platform Colorectal Cancer
Acronym: AZURITE
Status: Active, not recruiting | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-100452
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer Metastatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal Cancer Metastatic
  Interventions: Other: Physician's choice according to patient's needs.

INTERVENTIONS:
Other: Physician's choice according to patient's needs. — Routine care as per site standard.

SUMMARY:
The registry aims to collect and analyse information on the antineoplastic treatment of patients with metastatic colorectal cancer, treated in palliative intention in daily routine practice in Germany.

DETAILED DESCRIPTION:
AZURITE is a national, observational, prospective, longitudinal, multicenter cohort study (tumor registry platform) with the purpose to record information on the antineoplastic treatment of metastatic colorectal cancer in Germany. The registry will follow patients for up to three years. It will identify common therapeutic sequences and changes in the treatment of the disease. At inclusion, data in patient characteristics, comorbidities, tumor characteristics and previous treatments are collected. During the course of observation data on all systemic treatments, radiotherapies, surgeries, and outcome are documented.

Health-related quality of life (HRQoL) will be evaluated for up to three years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven metastatic colorectal cancer (stage IV) at time of inclusion (patients with metastatic disease and potential curative treatment intention are allowed)
* Age ≥ 18 years
* Planned first systemic therapy for metastatic disease
* Signed and dated informed consent form

  * Patients participating in the PRO module: prior to or at start of first systemic treatment for mCRC
  * Patients not participating in the PRO module: within four weeks after start of fist systemic therapy for mCRC

Exclusion Criteria:

* Patient who do not receive any systemic therapy for mCRC
* Patients whose metastatic disease was surgically resected prior to inclusion and who start adjuvant chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with metastatic (stage IV) colorectal cancer requiring palliative systemic first-line therapy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Course of treatment (treatment reality). | 3 years per patient.
  Documentation of anamnestic data and therapy sequences.

SECONDARY OUTCOMES:
Best Response. | 3 years per patient.
  Documentation of response rates per line of treatment.
Progression-free survival. | 3 years per patient.
  Documentation of progression-free survival per line of treatment.
Overall survival. | 3 years per patient.
  Documentation of overall survival per line of treatment.
Health-related quality of life (Patient-reported outcome, PRO). | 3 years per patient.
  EORTC QLQ-C30 core questionnaire [European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire; Scale 0-100; a high scale score represents a higher response level: (a) global health status: a high score represents high quality of life, (b) functional scales: a high score represents high/healthy level of functioning, (c) symptom scales/items: a high score represents high level of symptomatology or problems].
Carcinoma Health-related quality of life (Patient-reported outcome, PRO). | 3 years per patient.
  EORTC QLQ-CR29 [European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire; Scale 0-100; a high score for scales and single items represents a high level of symptomatology or problems].

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Graf, PD Dr., Study Chair — Deggendorf Institute of Technology, Faculty of Applied Healthcare Sciences; Frank Kullmann, Prof. Dr., Study Chair — Weiden i.d.O.; Marlies Michl, PD Dr., Study Chair — München; Jens Neumann, Prof. Dr., Study Chair — München; Roland Schnell, PD Dr., Study Chair — Frechen; Sebastian Stintzing, Prof. Dr., Study Chair — Berlin; Karin Potthoff, Dr., Study Chair — Freiburg i. Br.
Locations (1):
- Multiple sites all over germany, Multiple Locations, Germany